CLINICAL TRIAL: NCT01256671
Title: DHEA Against Vaginal Atrophy - Safety Study of 12 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC-230
Record Dates: First submitted 2010-12-03; First posted 2010-12-08 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Vaginal Atrophy
Keywords: Vulvar/Vaginal Atrophy; Atrophic Vaginitis; Dehydroepiandrosterone; DHEA; Prasterone; Vaginorm; Menopause; Intrarosa
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DHEA (Experimental): 0.5% DHEA (intravaginal)
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA — Vaginal suppository containing 0.5% (6.5 mg) DHEA; daily dosing with one suppository for 52 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone, Vaginorm

SUMMARY:
The purpose of this Phase III trial is to assess the long-term safety of intravaginal dehydroepiandrosterone (DHEA) in non-hysterectomized postmenopausal women with vaginal atrophy aged 40 to 75 years.

ELIGIBILITY:
Main Inclusion Criteria:

* Postmenopausal women (non-hysterectomized)
* Women between 40 and 75 years of age.
* Willing to participate in the study and sign an informed consent.
* Women who have self-identified symptom(s) of vaginal atrophy.
* Willing to have endometrial biopsy at screening and end of study (Week 52).

Main Exclusion Criteria:

* Undiagnosed abnormal genital bleeding.
* Hypertension equal to or above 140/90 mm Hg.
* The administration of any investigational drug within 30 days of screening visit.
* Endometrial hyperplasia, cancer or endometrial histology showing proliferative, secretory or menstrual type characteristics at histologic evaluation of endometrial biopsy performed at screening.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Principal Investigator — Clinical Research Center, Eastern Virginia Medical School, Norfolk, VA
Locations (41):
- United States (31):
  - EndoCeutics site # 39, Montgomery, Alabama
  - EndoCeutics site # 14, Tucson, Arizona
  - EndoCeutics site # 21, Sacramento, California
  - EndoCeutics site # 30, San Diego, California
  - EndoCeutics site # 17, San Diego, California
  - EndoCeutics site # 36, Denver, Colorado
  - EndoCeutics site # 42, Milford, Connecticut
  - EndoCeutics site # 07, Washington D.C., District of Columbia
  - EndoCeutics site # 45, Boynton Beach, Florida
  - EndoCeutics site # 26, Jacksonville, Florida
  - EndoCeutics site # 41, West Palm Beach, Florida
  - EndoCeutics site # 23, Sandy Springs, Georgia
  - EndoCeutics site # 10, Meridian, Idaho
  - EndoCeutics site # 27, Baltimore, Maryland
  - EndoCeutics site # 22, Kalamazoo, Michigan
  - EndoCeutics site # 25, Lincoln, Nebraska
  - EndoCeutics site # 24, Omaha, Nebraska
  - EndoCeutics site # 28, Moorestown, New Jersey
  - EndoCeutics site # 50, Neptune City, New Jersey
  - EndoCeutics site # 44, New Brunswick, New Jersey
  - EndoCeutics site # 19, New York, New York
  - EndoCeutics site # 16, Durham, North Carolina
  - EndoCeutics site # 33, Beachwood, Ohio
  - EndoCeutics site # 05, Cleveland, Ohio
  - EndoCeutics site # 47, Cleveland, Ohio
  - EndoCeutics site # 15, Columbus, Ohio
  - EndoCeutics site # 35, Pittsburgh, Pennsylvania
  - EndoCeutics site # 09, West Jordan, Utah
  - EndoCeutics site # 31, Charlottesville, Virginia
  - EndoCeutics site # 03, Norfolk, Virginia
  - EndoCeutics site # 38, Renton, Washington
- Canada (10):
  - EndoCeutics site # 13, Calgary, Alberta
  - EndoCeutics site # 06, Bathurst, New Brunswick
  - EndoCeutics site # 04, Drummondville, Quebec
  - EndoCeutics site # 34, Montreal, Quebec
  - EndoCeutics site # 12, Montreal, Quebec
  - EndoCeutics site # 02, Québec, Quebec
  - EndoCeutics site # 01, Québec, Quebec
  - EndoCeutics site # 18, Saint Romuald, Quebec
  - EndoCeutics site # 08, Shawinigan, Quebec
  - EndoCeutics site # 11, Sherbrooke, Quebec

REFERENCES:
- [Result] Labrie F, Archer DF, Bouchard C, Girard G, Ayotte N, Gallagher JC, Cusan L, Baron M, Blouin F, Waldbaum AS, Koltun W, Portman DJ, Cote I, Lavoie L, Beauregard A, Labrie C, Martel C, Balser J, Moyneur E; Members of the VVA Prasterone Group. Prasterone has parallel beneficial effects on the main symptoms of vulvovaginal atrophy: 52-week open-label study. Maturitas. 2015 May;81(1):46-56. doi: 10.1016/j.maturitas.2015.02.005. Epub 2015 Feb 16. PMID 25771041
- [Result] Bouchard C, Labrie F, Derogatis L, Girard G, Ayotte N, Gallagher J, Cusan L, Archer DF, Portman D, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Group. Effect of intravaginal dehydroepiandrosterone (DHEA) on the female sexual function in postmenopausal women: ERC-230 open-label study. Horm Mol Biol Clin Investig. 2016 Mar;25(3):181-90. doi: 10.1515/hmbci-2015-0044. PMID 26725467
- [Result] Ke Y, Gonthier R, Simard JN, Archer D, Lavoie L, Martel C, Vaillancourt M, Labrie F. Serum steroids remain within the same normal postmenopausal values during 12-month intravaginal 0.50% DHEA. Horm Mol Biol Clin Investig. 2015 Dec;24(3):117-29. doi: 10.1515/hmbci-2015-0035. PMID 26509785
- [Result] Portman DJ, Labrie F, Archer DF, Bouchard C, Cusan L, Girard G, Ayotte N, Koltun W, Blouin F, Young D, Wade A, Martel C, Dube R; other participating members of VVA Prasterone Group. Lack of effect of intravaginal dehydroepiandrosterone (DHEA, prasterone) on the endometrium in postmenopausal women. Menopause. 2015 Dec;22(12):1289-95. doi: 10.1097/GME.0000000000000470. PMID 25968836
- [Result] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 798 subjects were screened at 41 medical/research sites located in the US (31 centers) and Canada (10 centers) and 530 subjects were randomized. The first subject first visit was on 30-NOV-2010 and the last subject last visit was on 16-JUL-2012.
Groups:
- 0.50% DHEA: DHEA (prasterone): Vaginal suppository containing 0.50% (6.5 mg) DHEA; daily dosing with one suppository for 52 weeks.
Period: Overall Study
Arm/Group | 0.50% DHEA
Started | 530
Safety Population | 521
Completed | 435
Not Completed | 95
Not completed — Adverse Event | 29
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 31
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 4
Not completed — Non-compliance/Sponsor Decision/Other | 12

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population corresponds to the Safety Population which includes all subjects who received any amount of DHEA, and who have any safety information available.
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 521
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.95 (5.65)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 521
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Caucasian | 478
  Black or African American | 31
  Asian | 3
  American Indian or Alaska Native | 3
  Native Hawaiian or Other Pacific Islander | 2
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety of Intravaginal Prasterone (DHEA): Endometrium
Description: The long-term safety of intravaginal prasterone has been evaluated on different parameters including the endometrium. For this purpose, endometrial biopsies were performed at screening and at the end of the study (52 weeks) or at discontinuation visit for women who were exposed to intravaginal DHEA (prasterone) for at least 12 weeks. At screening, the endometrium had to be atrophic/inactive for women to be enrolled in the study. Only the end-of-study data are presented.
Time Frame: Baseline and Week 52 (or discontinuation)
Population: Only subjects in the Safety Population who had an end-of-study endometrial biopsy are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 457
Participants
  Endometrium: Atrophic/Inactive | 421
  Endometrium: No/Insufficient Tissue for Diagnosis | 36

2. Secondary Outcome: Change From Baseline to Week 52 of Vaginal Cell Maturation (Percentage of Parabasal Cells).
Description: The percentage of parabasal cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: Subgroups of the Safety Population were used for analysis. The subgroup identified "ALL" includes subjects meeting or not the vulvovaginal atrophy (VVA) criteria at Baseline while the subgroup "VVA" only includes subjects meeting VVA criteria (pH ˃5, superficial cells ≤ 5% and moderate/severe VVA symptom being most bothersome (MBS)).
Measure: Mean (Standard Error); unit: percentage of parabasal cells
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
percentage of parabasal cells
  Baseline: Subgroup ALL: number analyzed (Participants) | 454
  Baseline: Subgroup ALL | 55.49 (2.03)
  Week 52: Subgroup ALL: number analyzed (Participants) | 454
  Week 52: Subgroup ALL | 12.81 (0.97)
  Change from Baseline: Subgroup ALL: number analyzed (Participants) | 454
  Change from Baseline: Subgroup ALL | -42.67 (1.84)
  Baseline: Subgroup VVA: number analyzed (Participants) | 292
  Baseline: Subgroup VVA | 63.95 (2.41)
  Week 52: Subgroup VVA: number analyzed (Participants) | 292
  Week 52: Subgroup VVA | 14.80 (1.27)
  Change from Baseline: Subgroup VVA: number analyzed (Participants) | 292
  Change from Baseline: Subgroup VVA | -49.14 (2.22)

3. Secondary Outcome: Change From Baseline to Week 52 of Vaginal Cell Maturation (Percentage of Superficial Cells).
Description: The percentage of superficial cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of superficial cells
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
percentage of superficial cells
  Baseline: Subgroup ALL: number analyzed (Participants) | 454
  Baseline: Subgroup ALL | 2.02 (0.19)
  Week 52: Subgroup ALL: number analyzed (Participants) | 454
  Week 52: Subgroup ALL | 9.42 (0.36)
  Change from Baseline: Subgroup ALL: number analyzed (Participants) | 454
  Change from Baseline: Subgroup ALL | 7.41 (0.38)
  Baseline: Subgroup VVA: number analyzed (Participants) | 292
  Baseline: Subgroup VVA | 0.96 (0.08)
  Week 52: Subgroup VVA: number analyzed (Participants) | 292
  Week 52: Subgroup VVA | 8.81 (0.41)
  Change from Baseline: Subgroup VVA: number analyzed (Participants) | 292
  Change from Baseline: Subgroup VVA | 7.85 (0.42)

4. Secondary Outcome: Change From Baseline to Week 52 of Vaginal pH.
Description: A pH strip fixed on an Ayre spatula (or equivalent) was applied directly to the lateral wall of the vagina. The change in color of the pH indicator strip was compared to the color chart for pH evaluation. The corresponding pH value (with one decimal) was recorded. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: pH
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
pH
  Baseline: Subgroup ALL: number analyzed (Participants) | 457
  Baseline: Subgroup ALL | 6.23 (0.04)
  Week 52: Subgroup ALL: number analyzed (Participants) | 457
  Week 52: Subgroup ALL | 5.09 (0.04)
  Change from Baseline: Subgroup ALL: number analyzed (Participants) | 457
  Change from Baseline: Subgroup ALL | -1.14 (0.04)
  Baseline: Subgroup VVA: number analyzed (Participants) | 293
  Baseline: Subgroup VVA | 6.40 (0.04)
  Week 52: Subgroup VVA: number analyzed (Participants) | 293
  Week 52: Subgroup VVA | 5.13 (0.05)
  Change from Baseline: Subgroup VVA: number analyzed (Participants) | 293
  Change from Baseline: Subgroup VVA | -1.27 (0.05)

5. Secondary Outcome: Change From Baseline to Week 52 of Self-assessment of VVA Symptom Dyspareunia
Description: The severity of dyspareunia was evaluated by a questionnaire. The severity of dyspareunia recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: Overall, 476 subjects met vulvovaginal atrophy (VVA) criteria by having moderate/severe (MS) dyspareunia, dryness and/or irritation/itching. The analysis "MS" dyspareunia only includes subjects having MS dyspareunia (being or not most bothersome (MBS)) (n=240); the analysis "MBS/MS" only includes subjects with MS dyspareunia being MBS (n=183).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
units on a scale
  Baseline: Subgroup MS: number analyzed (Participants) | 240
  Baseline: Subgroup MS | 2.53 (0.03)
  Week 52: Subgroup MS: number analyzed (Participants) | 240
  Week 52: Subgroup MS | 0.85 (0.06)
  Change from Baseline: Subgroup MS: number analyzed (Participants) | 240
  Change from Baseline: Subgroup MS | -1.68 (0.06)
  Baseline: Subgroup MBS/MS: number analyzed (Participants) | 183
  Baseline: Subgroup MBS/MS | 2.57 (0.04)
  Week 52: Subgroup MBS/MS: number analyzed (Participants) | 183
  Week 52: Subgroup MBS/MS | 0.87 (0.07)
  Change from Baseline: Subgroup MBS/MS: number analyzed (Participants) | 183
  Change from Baseline: Subgroup MBS/MS | -1.69 (0.07)

6. Secondary Outcome: Change From Baseline to Week 52 of Self-assessment of VVA Symptom Vaginal Dryness
Description: The severity of vaginal dryness was evaluated by a questionnaire. The severity of vaginal dryness recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: Overall, 476 subjects met vulvovaginal atrophy (VVA) criteria by having moderate/severe (MS) dyspareunia, dryness and/or irritation/itching. The analysis "MS" only includes subjects having MS dryness (being or not most bothersome (MBS)) (n=251); the analysis "MBS/MS" only includes subjects with MS dryness being MBS (n=81).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
units on a scale
  Baseline: Subgroup MS: number analyzed (Participants) | 251
  Baseline: Subgroup MS | 2.22 (0.03)
  Week 52: Subgroup MS: number analyzed (Participants) | 251
  Week 52: Subgroup MS | 0.59 (0.05)
  Change from Baseline: Subgroup MS: number analyzed (Participants) | 251
  Change from Baseline: Subgroup MS | -1.63 (0.05)
  Baseline: Subgroup MBS/MS: number analyzed (Participants) | 81
  Baseline: Subgroup MBS/MS | 2.19 (0.04)
  Week 52: Subgroup MBS/MS: number analyzed (Participants) | 81
  Week 52: Subgroup MBS/MS | 0.67 (0.09)
  Change from Baseline: Subgroup MBS/MS: number analyzed (Participants) | 81
  Change from Baseline: Subgroup MBS/MS | -1.52 (0.09)

7. Secondary Outcome: Change From Baseline to Week 52 of Self-assessment of VVA Symptom Irritation/Itching
Description: The severity of irritation/itching was evaluated by a questionnaire. The severity of irritation/itching recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: Overall, 476 subjects met vulvovaginal atrophy (VVA) criteria by having moderate/severe (MS) dyspareunia, dryness and/or irritation/itching. The analysis "MS" only includes subjects having MS irritation/itching (being or not most bothersome (MBS)) (n=86); the analysis "MBS/MS" only includes subjects with MS irritation/itching being MBS (n=23).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 476
units on a scale
  Baseline: Subgroup MS: number analyzed (Participants) | 86
  Baseline: Subgroup MS | 2.10 (0.03)
  Week 52: Subgroup MS: number analyzed (Participants) | 86
  Week 52: Subgroup MS | 0.60 (0.08)
  Change from Baseline: Subgroup MS: number analyzed (Participants) | 86
  Change from Baseline: Subgroup MS | -1.50 (0.09)
  Baseline: Subgroup MBS/MS: number analyzed (Participants) | 23
  Baseline: Subgroup MBS/MS | 2.13 (0.07)
  Week 52: Subgroup MBS/MS: number analyzed (Participants) | 23
  Week 52: Subgroup MBS/MS | 0.74 (0.14)
  Change from Baseline: Subgroup MBS/MS: number analyzed (Participants) | 23
  Change from Baseline: Subgroup MBS/MS | -1.39 (0.16)

8. Primary Outcome: Long-term Safety of Intravaginal Prasterone (DHEA): Serum Steroid Levels
Description: The long-term safety of intravaginal prasterone has been evaluated on different parameters including the serum levels of DHEA and its metabolites. For this purpose, blood samples were collected at Baseline and different post-Baseline timepoints for the determination of serum steroid levels by a central laboratory using validated liquid chromatography tandem mass spectrometry (LC-MS/MS) methods. The serum levels of dehydroepiandrosterone (DHEA), estradiol (E2) and testosterone (TESTO) obtained at Baseline and Week 52 as well as the change from Baseline to Week 52 are presented.
Time Frame: Baseline and Week 52
Population: Data are presented for subjects in the Safety Population who have steroid data at both baseline and Week 52.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | 0.50% DHEA
Number analyzed (Participants) | 429
pg/mL
  DHEA: Baseline: number analyzed (Participants) | 426
  DHEA: Baseline | 2071.61 (65.70)
  DHEA: Week 52: number analyzed (Participants) | 426
  DHEA: Week 52 | 2997.25 (85.23)
  DHEA: Change from Baseline: number analyzed (Participants) | 426
  DHEA: Change from Baseline | 925.65 (74.35)
  E2: Baseline | 6.05 (1.11)
  E2: Week 52 | 4.46 (0.32)
  E2: Change from Baseline | -1.59 (1.13)
  TESTO: Baseline | 161.28 (6.93)
  TESTO: Week 52 | 189.44 (4.79)
  TESTO: Change from Baseline | 28.17 (6.55)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 52 (+ 30-day follow-up period after last dose)
Arm/Group | 0.50% DHEA
Serious Adverse Events (participants affected / at risk) | 18/521
Other Adverse Events (participants affected / at risk) | 177/521
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.50% DHEA (N=521)
Colitis ischaemic (Gastrointestinal disorders) | 1
Duodenal stenosis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Infectious peritonitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Cystocele repair (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Rectocele repair (Surgical and medical procedures) | 1
Arteriovenous fistula (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.50% DHEA (N=521)
Application site discharge (General disorders) | 73
Nasopharyngitis (Infections and infestations) | 51
Urinary tract infection (Infections and infestations) | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide to the SPONSOR 30 days prior to submission all documents for publication, presentation, etc that report any trial results. The SPONSOR shall have editorial rights on documents and the right to review/comment with regard to (1) proprietary information, (2) accuracy of the information, (3) correctness of the scientific evaluation/conclusions and (4) to ensure that the information is fairly balanced and in compliance with regulations.